CLINICAL TRIAL: NCT05520385
Title: Correlation Between Blood Group ,Rh and Obesity With Colorectal Carcinoma Among Patients Attending Al-kindy Teaching Hospital/Baghdad
Brief Title: Correlation Between Blood Group ,Rh and Obesity With Colorectal Carcinoma
Status: Completed | Type: Observational
Sponsor: Al-Kindy Teaching Hospital (Other)
Responsible Party: Principal Investigator, Safaa Hadi Abdulsattar Alshihmani, specialist doctor, Al-Kindy Teaching Hospital
Other Study IDs: colorectal CA
Record Dates: First submitted 2022-08-20; First posted 2022-08-29 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-09

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Blood Grouping and Crossmatching

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: blood group and Rh — check of blood group , Rh for patient and control

SUMMARY:
Aim of study: is there possibility of relationship between ABO blood group, Rh & obesity with CRC, that is what we tried to show in this study .

DETAILED DESCRIPTION:
Cancer is an important leading cause of great psychosocial and economic burden worldwide and about 1.23 million individual annually affected by CRC which is considered as the most common type of cancer ( 9.7 % of overall cancers )and 8 % ( 608,000 case ) died with CRC overall cancer death cases , so it's the fourth most common cause of death among different types of cancer .

There is variability in distribution of cases worldwide , as explained by epidemiological data which showed about 60 % of CRC cases presented in developed countries ( 2 % per year ) while in developing countries there is annual increase in the incidence of CRC cases with proportion occurring among patients with age ≤ 40 years is 2 - 8 percent in western countries while in middle east region its about 15 - 35 percent and the incidence rate is less in female than in male with favorable female gender as a prognostic factor over male .

There are three different risk groups for CRC, these are FAP, hereditary nonpolyposis colon cancer syndrome (lynch syndrome), and genetic mutations that lead to sporadic colon cancer .

The exact cause is unclear but many factors are involved including environmental and genetic . About 24 % of the cases with CRC are due to genetic factors while 75 % of the cases are sporadic and 1 % in patients with pre -existing IBD . Those who immigrates to area with high incidence of CRC from low incidence area may prone to develop CRC which may be related to consumption of red meat and decrease physical activity .

The environmental factors including dietary factors like : Lack of fiber , high-fat diet and exposure of mucosa to high levels of bile acids due to impairment of enterohepatic circulation which leading to form carcinogens from degradation of bile salts while previous cholecystectomy has not been proved to be risk for developing CRC .

Regarding genetic factors, there are several genes among them Tumor suppressor genes (e.g. APC, p53 ) , Oncogenes (e.g Ras) and Mismatch-repair genes (e.g hMSH2 and hMLH1) were identified as contributing to hereditary colorectal cancer .

Here in this study two factors will be discussed with their relation to development of CRC , those factors are ABO blood group , Rh factor and the other one is obesity and as following :

Actually , the first human genetic marker are antigens of the ABO system despite of they are a chemical component on erythrocyte membrane but showing expression on variety of epithelial cells including the mucosa of gastrointestinal tract, that was the leading cause observation studies on any correlation between ABO blood group , Rh with tumor .

From first studies, Aird et al in 1953 who reported a correlation between ABO Rh factor and carcinoma of stomach , also recently a significant association with pancreatic tumor had been reported . In addition to many studies showed a relationship between ABO antigen expression and CRC .

Regarding the obesity , about billion of people are now suffering from obesity worldwide which is considered as one of the strongest factors affecting many health conditions among them some cancers & the prevalence of obesity is rising in many Asian countries including Japan but still lower than western countries .

Many epidemiological studies identified high body mass index as independent risk factor for CRC , some of these studies in western countries showing a significant association between BMI and risk of CRC .

ELIGIBILITY:
Inclusion Criteria:

* patient with bleeding per rectum
* chronic pain in the right iliac fossa with anemia
* change in bowel habit
* constipation
* tinesmus .

Exclusion Criteria:

* Patient with history of other cancer
* those with chronic diseases like H.T, DM ,
* patients presenting with intestinal obstruction due to tumor
* athletics were excluded from the study

Ages: 30 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: those who attending Al-kindy Teaching Hospital for colonoscopic examination
Sampling Method: Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
an association between occurrence of CRC and blood group A+ , O + . | baseline
  Haemagglutination method was used to detect blood group and Rh factor for patients and control group

SECONDARY OUTCOMES:
an association between occurrence of CRC and overweight and class І obesity patients | basline
  Colonoscopy was done by using Olympus colonoscope , lucera CLV-260 and histopathological examination was done to confirm the diagnosis of CRC

CONTACTS AND LOCATIONS:
Overall Officials: Laith N. Hindoush, doctor, Study Chair — Baghdad/Iraq

IPD SHARING:
Plan to Share IPD: Undecided